CLINICAL TRIAL: NCT05982223
Title: Effectiveness of Integrative Medicine Treatments in Lymphoma Survivors
Brief Title: Integrative Medicine in Lymphoma Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0050-23-BNZ
Record Dates: First submitted 2023-07-16; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Lymphoma
Keywords: Lymphoma survivors; Integrative medicine; Complementary medicine; Quality of life; Shiatsu; Acupuncture; Hematology
MeSH Terms: conditions — Lymphoma | interventions — Acupuncture Therapy; Mind-Body Therapies; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Preference-based comparative effectiveness clinical trial
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative oncology (Experimental): All patients will be followed up by a haemato-oncologist. The frequency and type of visits and exams will be determined by National Comprehensive Cancer Network (NCCN) guidelines, patients' symptoms and physician's clinical judgement. Patients recruited to the intervention arm will receive, on top of the defined conventional medicine follow-up, integrative oncology intervention including emotional treatments (counseling, spiritual guidance), complementary medicine (acupuncture, herbal supplements, mind-body, touch and/or movement therapies) or both. The type and frequency of these interventions will be defined by the integrative team in coordination with the patient, based on evidence-based data, patient's symptoms, and preferences. The duration of the intervention will be 6 months from recruitment.
  Interventions: Procedure: Acupuncture; Procedure: Mind-body therapy; Procedure: Touch therapy; Procedure: Movement therapy; Dietary Supplement: Herbal supplements; Behavioral: Emotional treatment
- Conventional medicine only (No Intervention): All patients will be followed up by a haemato-oncologist. The frequency and type of visits and exams will be determined by NCCN guidelines, patients' symptoms and physician's clinical judgement.

INTERVENTIONS:
Procedure: Acupuncture — The frequency of acupuncture will be defined by the integrative team in coordination with the patient, based on evidence-based data, patient's symptoms, and preferences. The duration of the intervention will be 6 months from recruitment.
  Arms: Integrative oncology
Procedure: Mind-body therapy — The frequency of mind-body therapy (hypnosis, guided imagery) will be defined by the integrative team in coordination with the patient, based on evidence-based data, patient's symptoms, and preferences. The duration of the intervention will be 6 months from recruitment.
  Arms: Integrative oncology
Procedure: Touch therapy — The frequency of touch therapy (shiatsu, reflexology) will be defined by the integrative team in coordination with the patient, based on evidence-based data, patient's symptoms, and preferences. The duration of the intervention will be 6 months from recruitment.
  Arms: Integrative oncology
Procedure: Movement therapy — The frequency of movement therapy (Tai-Chi, Qi-Qong) will be defined by the integrative team in coordination with the patient, based on evidence-based data, patient's symptoms, and preferences. The duration of the intervention will be 6 months from recruitment.
  Arms: Integrative oncology
Dietary Supplement: Herbal supplements — The choice of herbal supplement will be defined by the integrative team in coordination with the patient, based on evidence-based data, patient's symptoms, and preferences. The duration of the intervention will be 6 months from recruitment.
  Arms: Integrative oncology
Behavioral: Emotional treatment — The frequency of emotional treatments (counseling, spiritual guidance) will be defined by the integrative team in coordination with the patient, based on evidence-based data, patient's symptoms, and preferences. The duration of the intervention will be 6 months from recruitment.
  Arms: Integrative oncology

SUMMARY:
Lymphoma is a cancer of the lymph nodes. While some are "silent" and only require follow-up, in cases of aggressive lymphoma, treatment is necessary, and usually includes biological drugs, chemotherapy or both. These drugs often cause significant damage to quality-of-life and various symptoms that do not always go away. Although the treatments are often limited in time and with recovery rates over 60%, most patients are left with a significantly impaired quality-of-life and difficulty in returning to their previous life. Many studies, most of which were conducted in breast cancer survivors, show the place of complementary medicine in the recovery process, both in terms of symptom relief and in improving quality-of-life. Few studies have examined the place of complementary and integrative medicine in lymphoma survivors. The purpose of the present study is to examine the effect of integrative treatments (a combination of conventional and complementary medicine) on quality-of-life of lymphoma survivors, on specific symptoms caused by the disease and its treatment, on economic and social aspects, as well as on the course of the disease. At the hematological unit of Bnai Zion Medical Center, Haifa, Israel, patients with lymphoma who have received chemotherapy, biological treatment or both, and have been defined as recovering by the treating hematologist, will be offered a choice of different types of complementary medicine (acupuncture, herbal medicine, mind-body, movement and touch therapies), emotional treatment (conversations with social worker, spiritual guidance), or both, in addition to the medical and nursing care offered to all survivors. Patients who prefer not to come to the clinic for these treatments will be assigned to the control group and will fill out questionnaires only. The duration of the treatments will be six months and follow-up for another two years. The type of treatments the patient will receive will be chosen in coordination between the integrative team and the patient and according to the symptoms. An assessment will be made on the effect of these treatments on quality-of-life of lymphoma survivors (based on questionnaires), including physical, psycho-spiritual and economic aspects, as well as on the course of the disease.

DETAILED DESCRIPTION:
Background: Lymphoma is a malignant disease of the lymph nodes. While some of the lymphomas are indolent and require only follow-up, in cases of aggressive lymphoma or indolent lymphoma with a high burden of disease, treatment is necessary and usually includes biological drugs, chemotherapy or both. These drugs often cause significant damage to quality-of-life, including various symptoms such as fatigue, gastrointestinal symptoms, neuropathy, as well as psycho-emotional and financial damage surrounding the cessation of work during the treatments. Although the treatments are often limited in time and with recovery rates above 60% in the case of aggressive lymphoma, most patients are left with a significant impairment in the quality-of-life and difficulty in returning to the life before the disease. Survivor clinics are usually located outside the oncology clinics and are designed to help cancer patients return to life after they have recovered from the disease. Many studies, mostly in breast cancer survivors, show the place of complementary medicine in the recovery process, both in terms of relieving symptoms and improving quality-of-life. Few studies have examined the place of complementary medicine in survivor clinics in haemato-oncological patients after intensive and time-limited treatments. In addition, integrative oncology that incorporates both conventional and complementary medicine, is a developing discipline that has been shown to be effective in the relief of many cancer-related symptoms such as chemotherapy-induced peripheral neuropathy, which is common in lymphoma survivors, and other outcomes such as quality-of-life, or even survival.

Hypothesis: In the present study, we assumed that an integrative oncology approach was effective for improving different outcomes of lymphoma survivors including quality-of-life, specific symptoms caused by the disease and its treatment, economic and social aspects, as well as the course of the disease.

Study plan: At the Hematology Unit at Bnai Zion Hospital, adult lymphoma survivors that received chemotherapy, biologic therapy or both during active lymphoma treatment, and are willing to participate in the study, will be recruited up to one year after remission. After completing questionnaires and an initial assessment by the integrative team, the patients will be divided by preference between the control group who will receive the mandatory basic treatment for follow-up after the disease (medical and nursing); and the intervention group who will come to the clinic and receive, in addition to the above, emotional treatments (counseling, spiritual guidance), complementary medicine (acupuncture, herbal supplements, mind-body, touch and/or movement therapies) or both. The type and frequency of complementary therapy will be chosen by the integrative team in coordination with the patient, based on patient's symptoms and preferences. The duration of the intervention will be 6 months from recruitment. During follow-up, the patients will fill-out a MYCAW questionnaire to assess symptoms in each treatment (or once a month in the control group) and a safety assessment will be performed using the validated Acupuncture-Adverse Events (Acup-AE) questionnaire for acupuncture or targeted questioning for other treatments. Also, the patients will fill-out quality-of-life questionnaires once a month and economic and cognitive evaluation questionnaires once every 3 months. The haemato-oncologist will complete an assessment of the disease state once every 3 months. In addition, 3 months after the end of the treatments, the patients will fill-out all the same questionnaires for follow-up. The haemato-oncologist will perform a medical follow-up on the condition of the disease once every 3 months for two years from the end of the treatments at the survivor clinic.

The primary outcome is the effect of an integrative approach on quality-of-life of lymphoma survivors. Secondary outcomes include the effect of such approach on specific symptoms caused by the disease and its treatment, economic and social aspects, as well as on the course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a lymphoproliferative disease
* Aged 18 years or older
* Received chemotherapy, biological treatment or both for treating the lymphoproliferative disease
* Defined in remission for less than one year by the haemato-oncologist (maintenance therapy is authorized)
* Can respond to questionnaires
* Signed informed consent

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Quality-of-life by EQ-5D scale | Through study completion: an average of 1 year
  EQ-5D scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient indicates health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ visual analogue scale (VAS) records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.

SECONDARY OUTCOMES:
Symptom relief | Through study completion: an average of 1 year
  Measure Yourself Concerns and Wellbeing (MYCAW) questionnaire: requires participants to nominate one or two concerns and, using a seven-point scale from 0 (worse outcome) to 6 (best outcome), to score these concerns and their general feeling of wellbeing
Cognitive functions | Through study completion: an average of 1 year
  Functional Assessment of Cancer Therapy - cognitive (FACT-cog) questionnaire: evaluates perceived cognitive functioning and their impact on quality of life. This is a self-reported 37-item questionnaire that consists of four subscales: Perceived Cognitive Impairment (CogPCI) (20 items), Perceived Cognitive Ability (CogPCA) (9 items), Comments from Others on Cognitive Function (Cog-Oth) (4 items), and Impact on Quality of Life (Cog-QoL) (4 items). All items are rated for the previous week, including the day of administration, on a 5-point Likert scale ranging from 0 "Never" or "Not at all" to 4 "Several times a day" or "Very much". The total CogPCI subscale ranges from 0 to 72, the CogPCA ranges between 0 and 28, and each of the Cog-QoL and Cog-Oth ranges between 0 and 16. The total score for the FACT-Cog is computed by summing all the item scores and ranges from 0 to 148 points, with a higher score indicative of better perceived cognitive functioning.
Perception of disease control | Through study completion: an average of 1 year
  Perceived Personal Control (PPC) scale: a 4-questions-scale, with each question evaluating in a 0-4 scale the perception of disease control (0: worse control to 4: best control)
Economic evaluation | Through study completion: an average of 1 year
  Questionnaire on the measurement, valuation, and estimation of costs adapted from a validated questionnaire on informal care
Adverse events | Through study completion: an average of 1 year
  A checklist with acupuncture adverse events based on the Acupuncture-Adverse Events (AcupAE) questionnaire will be used to evaluate acupuncture-associated safety events after each treatment. For non-acupuncture complementary medicine therapies, the practitioner will directly question and evaluate the patient after each intervention for possible safety events. Specifically for dietary and herbal supplements, adverse events and interactions will be evaluated at each visit, and the Naranjo and adapted Drug Interaction Probability Scales (DIPS) will be used to assess the causality of such events with the specific dietary supplements.
Relapse of lymphoma | 3 years
  Based on clinical evaluation of the physician
Progression-free survival | 3 years
  Time from screening to the occurrence of disease progression or death, based on clinical evaluation
Overall survival | 3 years
  Time from screening to death, based on clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Levy Yurkovski, MD, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT05982223/Prot_SAP_000.pdf